CLINICAL TRIAL: NCT02152020
Title: Patient-Centered Integration of Acupuncture to Decrease Pain for Cancer Survivors
Brief Title: Patient-Centered Acupuncture for Pain (PCAP)
Status: Completed | Type: Observational
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: UPCC 01914
Record Dates: First submitted 2014-05-29; First posted 2014-06-02 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: Cancer Survivors
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Cancer survivors
  Interventions: Behavioral: Survey

INTERVENTIONS:
Behavioral: Survey

SUMMARY:
The objective of this study is to find out if acupuncture can improve the management of pain in cancer patients when used as part of a treatment plan that includes conventional pain medications. The investigators will enroll 36 cancer patients at Abramson Cancer Center and Penn Cancer Network sites. Participants will be enrolled in either the Conventional Pain Management group or Integrative Pain Management group.

ELIGIBILITY:
Inclusion Criteria:

* Women or men age 18 years or older
* Primary diagnosis of cancer with history of stage I, II, or III cancer
* Finished primary cancer treatments (surgery, chemotherapy, radiotherapy)
* Have a Karnofsky score of 60 or greater
* Can understand written English
* Have worst pain rated at least 4 or greater on an 11-point (0-10) numerical rating scale in the preceding week
* Have been taking pain medications daily
* Have had at least 15 days with pain in the preceding 30 days.

Exclusion Criteria:

* Women or men with metastatic (stage IV) cancer
* Unstable and progressive medical conditions as judged by the PIs or designated research nurse at the community hospitals (e.g., progressive cancer, uncontrolled heart failure) that may require hospitalization in the next 12 weeks
* Planned surgical procedures in the next 12 weeks
* Patients currently in a pain crisis as judged by the PI or designated research nurse that may warrant acute titration of medications or hospitalization
* Women who are pregnant or breastfeeding
* Unwillingness to adhere to study related procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer survivors 18 years or older with pain ratings of 4 or greater on a 0-10 numerical rating scale; primary diagnosis of cancer (stages I-III); finished primary cancer treatment; Karnofsky score 60 or greater; and who have been taking pain medications daily.
Sampling Method: Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2014-05; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Events | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jun Mao, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States